CLINICAL TRIAL: NCT06940518
Title: Phase II Trial of Ivonescimab in Previously Treated Patients With Advanced Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Strategic Alliance (Unknown); Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0277; NCI-2025-02811 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Ivonescimab; Clear Cell Renal Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 2 - (Post-ICB/VEGFTKI) (Experimental): Treatment with Ivonescimab IV Q3W
  Interventions: Drug: Ivonescimab
- Cohort 1 - (Post-pure-ICB) (Experimental): Treatment with Ivonescimab IV Q3W
  Interventions: Drug: Ivonescimab

INTERVENTIONS:
Drug: Ivonescimab — Given by IV

SUMMARY:
To learn if ivonescimab can help to control previously treated, locally advanced or metastatic ccRCC.

DETAILED DESCRIPTION:
Primary Objectives To determine the efficacy of objective response rate (ORR) and 24-week disease control rate (DCR), per RECIST 1.1, of ivonescimab monotherapy in participants with locally advanced or metastatic renal cell carcinoma with a clear cell component who had progression on at least one prior line of therapy.

Secondary Objectives To determine the safety profile of ivonescimab monotherapy in patients with locally advanced or metastatic renal cell carcinoma with a clear cell component who had progression on at least one prior line of therapy. To determine the overall survival (OS), progression free survival (PFS), duration of response (DOR), and adverse events with ivonescimab monotherapy in patients with locally advanced or metastatic renal cell carcinoma with a clear cell component who had progression on at least one prior line of therapy.

ELIGIBILITY:
Inclusion Criteria

1. Participants with histologically or cytologically confirmed metastatic/advanced clear cell RCC with a clear cell component who have received at least one prior line of systemic treatment in the advanced or metastatic setting, including a PD-1/PD-L1 checkpoint inhibitor administered in metastatic/advanced setting.

   1. Participants in cohort 1 must have not received a treatment containing a VEGF- or HIF2a(- directed agent in prior treatment lines of treatment for metastatic/advanced RCC
   2. Participants in cohort 2 must have had progression on or after at least one prior line of treatment containing a VEGF-directed agent in prior lines of therapy
2. Participants must have had evidence of disease progression on or after last treatment regimen received.
3. Participants who received HIF-2ƒ¿ inhibitors in prior lines of therapy are eligible in cohort 2 but not cohort 1.
4. Participants who received adjuvant immune checkpoint inhibitor are eligible, provided that they had progression while on adjuvant therapy, in which case they would be enrolled in cohort 1. Participants who recur after completing adjuvant therapy should receive a PD-1/PD-L1 checkpoint inhibitor in the advanced/metastatic setting to be eligible.
5. Participants must have at least one measurable site of disease per RECIST version 1.1. This is defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). For non-lymph node tumor lesions, they must be a minimum size of ≥ 10 mm. For malignant lymph node lesions, they must be at least ≥ 15 mm in short axis with conventional techniques or ≥10 mm with more sensitive techniques such as MRI or spiral CT scan. If the participant has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
6. ECOG performance status ≤2
7. Age ≥ 18 years
8. Participants must have adequate organ and marrow function prior to study entry as defined below:
9. INR and PT ≤ 1.5 x ULN and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤1.5 ULN (unless abnormalities are unrelated to coagulopathy). Therapeutic anticoagulation is permitted if: on a stable dose of low molecular weight heparin (LMWH) for > 2 weeks (14 days) at the time of enrollment or on a direct oral anticoagulant (DOAC) for > 2 weeks at time of enrollment.
10. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
11. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
12. Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. Patients who are Hepatitis C virus antibody positive (HCV Ab

    +) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
13. Participants with a history of major psychiatric illness must be judged (by the treating physician) able to fully understand the investigational nature of the study and the risks associated with the therapy.
14. The effects of Ivonescimab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy

    # CLN1114). This includes all female participants , between the onset of menses (as early as 8years of age) and 55 years unless the participants presents with an applicable exclusionary factor which may be one of the following: i. Postmenopausal (no menses in greater than or equal to 12 consecutive months). ii. History of hysterectomy or bilateral salpingo-oophorectomy. iii. Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy). iv. History of bilateral tubal ligation or another surgical sterilization procedure.
15. Female participants of childbearing potential (not postmenopausal for at least 12 months and not surgically sterile) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) before study entry. Pregnancy test must be repeated on the day of first infusion, if test performed > 14 days before starting study drug.
16. Female participants of childbearing potential having sex with an unsterilized male partner must agree to use a highly effective method of contraception from the beginning of screening until 90 days after the last dose of the ivonescimab. Unsterilized male patients having sex with a female partner of childbearing potential, or a pregnant or breastfeeding partner must agree to use barrier contraception (male condom) for the duration of the treatment period until 90 days after the last dose of ivonescimab. Male patients with female partners of childbearing potential must have the female partner agree to use at least 1 form of highly effective contraception for the duration of the treatment period until 90 days after the last dose of ivonescimab.

    1. Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

       * Ability to understand and the willingness to sign a written informed consent document for this clinical trial and the companion Trials LAB02-152 and PA17-0577

Exclusion Criteria:

1. Participants must not have any other malignancies within the past 2 years except for in situ carcinoma of any site, or adequately treated (without recurrence post-resection or postradiotherapy) carcinoma of the cervix or basal or squamous cell carcinomas of the skin, ductal carcinoma in situ of the breast or low-risk early stage prostate adenocarcinoma with negligible risk of metastasis or death.
2. Major surgical procedures or serious trauma within 4 weeks prior to enrollment, or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to enrollment.
3. Current hypertension with systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg after adequate oral antihypertensive therapy.
4. History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to enrollment, including but not limited to:

   o Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots).

   Transient hemoptysis associated with diagnostic bronchoscopy is allowed.
   * Nasal bleeding /epistaxis. Bloody nasal discharge is allowed.
   * Hematuria associated with urinary obstruction. Microhematuria or macrohematuria not associated with urinary obstruction are allowed.
   * Radiologically documented evidence of major blood vessel encasement with narrowing of the vessel that the investigator determines will pose a significantly increased risk of bleeding.
5. History of major diseases prior to enrollment, specifically:

   * Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification . grade 2) or vascular disease (eg, aortic aneurysm at risk of rupture) that required hospitalization within 12 months prior to randomization, or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
   * History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months prior to enrollment.
6. History of arterial thromboembolic event, venous thromboembolic event of Grade 3 and above as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 12 months prior to enrollment.

   * Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks prior to enrollment.
   * History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to enrollment.
7. Symptomatic CNS metastases, leptomeningeal disease, CNS metastases with hemorrhagic features, CNS metastasis ≥ 1.5 cm, CNS radiation within 7 days prior to enrolmment, or potential need for CNS radiation within the first cycle of ivonescimab.

   o Participants with treated/stable brain metastases are allowed on protocol if they had brain metastases that received CNS-directed therapy, such as surgery or treatment with radiosurgery or Gamma knife, without recurrence or edema for at least 1 month (4 weeks). Participants actively requiring glucocorticoids for uncontrolled brain or leptomeningeal metastases are not eligible. Participants must have stopped corticosteroids or be on physiologic corticosteroid replacement therapy (prednisone . 10 mg daily or equivalent).
8. Active or prior history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic inflammatory diarrhea).
9. Participants who are receiving any other investigational agents.
10. Active autoimmune disease requiring systemic therapy (e.g., with disease modifying drugs, prednisone >10 mg daily or equivalent, immunosuppressant therapy) within 2 years prior to enrollment. However the following will be allowed:

    * Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is permitted.
    * Intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections is permitted.
11. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
12. Severe infection within 4 weeks prior to enrollment, including but not limited to comorbidities requiring hospitalization, severe sepsis, or severe pneumonia; active infection (as determined by the investigator) requiring systemic anti-infective therapy within 2 weeks prior to enrollment (excluding antiviral therapy for hepatitis B or C).
13. Uncontrolled pleural effusions, pericardial effusions, or ascites that is clinically symptomatic. Participants managed with indwelling catheters (e.g., PleurX) are allowed.
14. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ivonescimab or other agents used in study. This includes known history of severe hypersensitivity to other monoclonal antibodies.
15. Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
16. Participants with active hepatitis B are required to have stable or declining levels of hepatitis B DNA by polymerase chain reaction (PCR) on appropriate anti-viral therapy with acceptable tolerability for one month prior to enrollment. All patients with active hepatitis C (hepatitis C virus [HCV] antibody positive with HCV RNA levels above the lower limit of detection) are excluded.
17. Pre-existing peripheral neuropathy that is ≥ Grade 2 by CTCAE version 5.0.
18. Pregnant women are excluded from this study because ivonescimab is a bispecific agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ivonescimab, breastfeeding should be discontinued if the mother is treated with ivonescimab.

    These potential risks may also apply to other agents used in this study.
19. Participant is breastfeeding or plans to breastfeed during the study.
20. Participants with persistent grade ≥ 2 adverse events per NCI CTCAE v5.0 from prior systemic therapies that would confound timely detection of immune-related adverse events due to ivonescimab or otherwise hinder patient participation in the clinical trial.
21. History or current evidence of any condition (medical [including adverse events from prior anticancer therapy, disorders secondary to tumor], surgical or psychiatric [including substance abuse]), or laboratory abnormality that might confound the results of the study, interfere with the participants participation for the full duration of the study, might lead to higher medical risk and/or is not in the best interest of the patient to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2028-01-19 (Estimated); Study Completion 2030-01-19 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version

CONTACTS AND LOCATIONS:
Overall Officials: Pavlos Msaouel, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org